CLINICAL TRIAL: NCT02674581
Title: An Open-label Study to Evaluate the Pharmacokinetics and Safety of BMS-663068 in Subjects With Normal Renal Function and Subjects With Mild, Moderate, Severe, and End-Stage Renal Dysfunction
Brief Title: A Study of the Pharmacokinetics and Safety of BMS-663068 Administered in Subjects With Normal Renal Function and With Mild, Moderate, Severe and End Stage Renal Dysfunction (ESRD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 206217; AI438-070 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2015-12-21; First posted 2016-02-04 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — fostemsavir; Prodrugs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Healthy Subjects (Experimental): A single dose of pro-drug, BMS-663068, administered orally and then metabolized to active BMS-626529 on Day 1.
  Interventions: Drug: Oral BMS-663068 (pro-drug)
- Mild Renal Impairment Subjects (Experimental): A single dose of pro-drug, BMS-663068, administered orally and then metabolized to active BMS-626529 on Day 1.
  Interventions: Drug: Oral BMS-663068 (pro-drug)
- Moderate Renal Impairment Subjects (Experimental): A single dose of pro-drug, BMS-663068, administered orally and then metabolized to active BMS-626529 on Day 1.
  Interventions: Drug: Oral BMS-663068 (pro-drug)
- Severe Renal Impairment Subjects (Experimental): A single dose of pro-drug, BMS-663068, administered orally and then metabolized to active BMS-626529 on Day 1.
  Interventions: Drug: Oral BMS-663068 (pro-drug)
- End Stage Renal Disease Subjects (Experimental): A single dose of pro-drug, BMS-663068, administered orally and then metabolized to active BMS-626529 on Day 1.
  Interventions: Drug: Oral BMS-663068 (pro-drug)

INTERVENTIONS:
Drug: Oral BMS-663068 (pro-drug) — Oral BMS-663068 (pro-drug), metabolized to active BMS-626529

SUMMARY:
An oral dose in healthy and renally impaired subjects to determine the drug effect for BMS-663068.

ELIGIBILITY:
Inclusion Criteria (For renal impaired subjects):

* Classification by renal function based on eGFR
* Clinical, ECG, and laboratory findings consistent with renal dysfunction
* BMI of 18.0 to 38.0 kg/m2 inclusive
* Women of child bearing potential (WOCBP) and sexually active fertile men with partners who are WOCBP must use non-hormonal highly effective birth control
* Slightly different inclusion criteria are defined in the protocol for healthy subjects

Exclusion Criteria:

* History of uncontrolled or unstable cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematopoietic, psychiatric, and/or neurological disease within 6 months of screening
* Evidence of rapidly deteriorating renal function, defined as a screening eGFR that has decreased from a previous eGFR by ≥ 50% within the last 3 months
* Current or recent (within 3 months of study drug administration) clinically significant gastrointestinal disease or gastrointestinal surgery (including cholecystectomy) that could impact the absorption of study drug
* Any major surgery within 4 weeks of study drug administration.
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02-26 (Actual); Primary Completion 2016-05-24 (Actual); Study Completion 2016-05-24 (Actual)

PRIMARY OUTCOMES:
Effect of Renal Impairment on The Primary Endpoints of Cmax | Day 1 - Day 5
  To assess the effect of varying degrees of renal impairment on the exposure of BMS-626529 after a single oral-dose administration of the pro-drug, BMS-663068, will be evaluated by assessing the primary endpoints of Cmax, for BMS-626529.

SECONDARY OUTCOMES:
Safety and Tolerability as assessed by the Incidence of Serious Adverse Events (SAEs), Adverse Events (AEs), AEs leading to discontinuation, and the results of ECGs, vital signs, physical examination, and clinical laboratory tests. | Day 1 - Day 5
  To assess the safety and tolerability of BMS-663068 in subjects with normal renal function and subjects with impaired renal functions, will be measured by the following secondary endpoints: Incidence of AEs, Serious Adverse Events (SAEs), and AEs leading to discontinuation, and results of vital signs, ECGs, physical examination, and clinical laboratory tests.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Miami, Florida, United States